CLINICAL TRIAL: NCT04209049
Title: An Open-label Trial Investigating the Pharmacokinetics and the Tolerability of NNC0174-0833 in Subjects With Normal Renal Function and Impaired Renal Function
Brief Title: A Research Study Looking Into Blood Levels of NNC0174-0833 in People With Normal and Impaired Kidney Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN9838-4518; U1111-1228-9001 (Other: World Health Organization (WHO))
Record Dates: First submitted 2019-12-19; First posted 2019-12-23 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Normal renal function (Experimental): All subjects will receive one dose of NNC0174-0833.
  Interventions: Drug: NNC0174-0833
- Mild renal impairment (Experimental): All subjects will receive one dose of NNC0174-0833.
  Interventions: Drug: NNC0174-0833
- Moderate renal impairment (Experimental): All subjects will receive one dose of NNC0174-0833.
  Interventions: Drug: NNC0174-0833
- Severe renal impairment (Experimental): All subjects will receive one dose of NNC0174-0833.
  Interventions: Drug: NNC0174-0833

INTERVENTIONS:
Drug: NNC0174-0833 — A single subcutaneous (s.c., under the skin) dose of 0.6 mg NNC0174-0833.

SUMMARY:
The study looks at the blood levels of a new study medicine in people with normal and impaired kidney function. Participants will get the study medicine called NNC0174-0833. This is an experimental medicine and has not been approved by the US FDA. It is being developed as a new medicine for weight management. Participants will get 1 injection of the study medicine by a study nurse at the clinic. The injection will be with a needle in a skin fold in the stomach area. The study will last for about 9 weeks. Participants will have about 7 visits with the study staff or the doctor. At the visits, participants will have clinical checks done and blood samples taken. Participants will be collecting their urine several times during the study. Participants will be asked about their health, medical history and habits. People who are already in another research study cannot take part. Only women who are not able to become pregnant can take part in the study. Only men who do not plan to father a child during the study or 6 weeks following the dose administration can take part in the study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female of non-childbearing potential, aged 18-80 years (both inclusive) at the time of signing informed consent.
* Meeting the pre-defined GFR criteria using estimated GFR (eGFR) based on serum creatinine for any of the renal function groups:
* For subjects with normal renal function: eGFR of equal to or above 90 mL/min
* For patients with mild renal impairment: eGFR of 60-89 mL/min
* For patients with moderate renal impairment: eGFR of 30-59 mL/min
* For patients with severe renal impairment: eGFR of <30 mL/min not requiring dialysis

Exclusion Criteria:

* Any disorder, which in the investigator's opinion might jeopardise subject's safety or compliance with the protocol.
* Use of prescription or non-prescription drugs, or non-routine vitamins, which at the investigators judgement may affect subject safety or the results of the trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2021-01-05 (Actual); Study Completion 2021-01-05 (Actual)

PRIMARY OUTCOMES:
Area under the plasma NNC0174-0833 concentration-time curve after a single dose | From baseline (Visit 2, Day 1, pre-dose) until completion of the end of trial visit (Visit 7, Day 36)
  nmol*h/L

SECONDARY OUTCOMES:
Maximum observed plasma NNC0174-0833 concentration after a single dose | From baseline (Visit 2, Day 1, pre-dose) until completion of the end of trial visit (visit 7, Day 36)
  nmol/L
Time to maximum observed plasma NNC0174-0833 concentration after a single dose | From baseline (Visit 2, Day 1, pre-dose) until completion of the end of trial visit (Visit 7, Day 36)
  hours
Number of treatment emergent adverse events (TEAEs) | From time of trial product administration (Visit 2, Day 1) until completion of the end of trial visit (Visit 7, Day 36)
  Number of events

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure (1452), Study Director — Novo Nordisk A/S
Locations (2):
- United States (2):
  - Novo Nordisk Investigational Site, Miami, Florida
  - Novo Nordisk Investigational Site, Orlando, Florida

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com